CLINICAL TRIAL: NCT00419952
Title: A 52-week, Randomised, Double-blind, Parallel-group, Multi-centre, Phase IIIB Study Comparing the Long Term Safety of SYMBICORT® pMDI 160/4.5 mg x 2 Actuations Twice Daily to Budesonide HFA pMDI 160 mg x 2 Actuations Twice Daily in Adult/Adolescent (≥12 Years) African American Subjects With Asthma
Brief Title: A Comparison of SYMBICORT® pMDI With Budesonide HFA pMDI in African American Subjects With Asthma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5896C00022
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-09

CONDITIONS: Asthma
Keywords: Moderate Asthma; Severe Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Symbicort (Experimental): Symbicort pMDI 160/4.5 ug x 2 actuations twice daily (BID)
  Interventions: Drug: Budesonide/formoterol (SYMBICORT) pMDI
- Budesonide (Experimental): Budesonide HFA pMDI 160 ug x 2 actuations BID
  Interventions: Drug: Budesonide HFA pMDI

INTERVENTIONS:
Drug: Budesonide/formoterol (SYMBICORT) pMDI — Symbicort pMDI 160/4.5 ug x 2 actuations twice daily (BID)
  Arms: Symbicort
Drug: Budesonide HFA pMDI — Budesonide HFA pMDI 160 ug x 2 actuations BID
  Arms: Budesonide

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of SYMBICORT® pMDI (a medication approved by the Food and Drug Administration, FDA) in the African American population.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, African American (self-reported), ≥12 years of age
* Moderate to severe asthma requiring treatment with an inhaled corticosteroid
* Diagnosis of asthma for at least 6 months

Exclusion Criteria:

* Subjects requiring treatment with systemic corticosteroids (e.g., oral, parenteral, ocular)
* Any significant disease or disorder that may jeopardize a subject's safety

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christer Hultquist, MD, Study Director — AstraZeneca
Locations (122):
- United States (122):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Muscle Shoals, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Buena Park, California
  - Research Site, Foothill Ranch, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Riverside, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, San Diego, California
  - Research Site, Stockton, California
  - Research Site, Torrance, California
  - Research Site, Winnetka, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Altamonte Springs, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Destin, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, Opa-locka, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, South Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Albany, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Stone Mountain, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, River Forest, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Merrillville, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Owensboro, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Bogalusa, Louisiana
  - Research Site, Marrero, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Sunset, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Mitchellville, Maryland
  - Research Site, Montgomery Village, Maryland
  - Research Site, Wheaton, Maryland
  - Research Site, Russells Mills, Massachusetts
  - Research Site, Bay City, Michigan
  - Research Site, Paw Paw, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Prentiss, Mississippi
  - Research Site, Vicksburg, Mississippi
  - Research Site, Omaha, Nebraska
  - Research Site, Blackwood, New Jersey
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Verona, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Newburgh, New York
  - Research Site, North Syracuse, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Tonawanda, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Highpoint, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Lyndhurst, Ohio
  - Research Site, Parma, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Beaver, Pennsylvania
  - Research Site, Collegeville, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Havertown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, Yardley, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Killeen, Texas
  - Research Site, Missouri City, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Sugarland, Texas
  - Research Site, Waco, Texas
  - Research Site, Hampton, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Springfield, Virginia

REFERENCES:
- See also: Related Info — http://www.asthmaclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 8 February 2007, the last patient completed the study on 30 November 2009. The study randomized participants only in the United States.
Pre-assignment Details: The study included a run-in period of 2 weeks when all patients were prescribed budesonide HFA pMDI 160 μg times 2 actuations BID at individual daily doses and rescue medication, as needed. To be randomized to treatment the patients needed to show pre-dose FEV1 of ≥50%. One patient in the budesonide group did not receive any dose.
Groups:
- Symbicort: Symbicort pMDI 160/4.5 ug x 2 actuations (twice daily) BID
- Budesonide: Budesonide HFA pMDI 160 ug x 2 actuations (twice daily) BID
Period: Overall Study
Arm/Group | Symbicort | Budesonide
Started | 377 | 365
Completed | 228 | 240
Not Completed | 149 | 125
Not completed — Adverse Event | 8 | 10
Not completed — Withdrawal by Subject | 44 | 43
Not completed — Lost to Follow-up | 43 | 34
Not completed — Protocol Violation | 32 | 24
Not completed — Pregnancy | 4 | 2
Not completed — Physician Decision | 1 | 3
Not completed — Incorrectly enrolled | 10 | 3
Not completed — Intake of prohibited medication | 2 | 2
Not completed — Occurence of 2 or more exacerbations | 2 | 0
Not completed — Diary or medication non-compliance | 2 | 4
Not completed — Abnormal ECG | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort | Budesonide | Total
Number analyzed (Participants) | 377 | 365 | 742
Age Continuous [Mean (Standard Deviation); unit: Years] | 36.19 (15.67) | 38.35 (15.22) | 37.27 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 232 | 481
  Male | 128 | 133 | 261

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Asthma Exacerbations
Description: An exacerbation was defined as symptomatic worsening requiring oral/systemic glucocorticoid therapy and/or emergency room visit and/or urgent care center visit and/or hospitalization.
Time Frame: 52 Weeks
Population: The full analysis set, consisting of all randomized patients who received at least one dose of randomized study medication and for whom data were collected after randomization.
Measure: Number; unit: Exacerbations
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 377 | 364
Exacerbations | 36 (NA) | 61 (NA)

2. Secondary Outcome: Asthma Exacerbations
Description: Number of participants with at least 1 exacerbation
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 377 | 364
Participants | 29 [-1.01 to 0.79] | 51 [-1.23 to 0.61]

3. Secondary Outcome: QT Interval Corrected Using the Fridericia Formula Measured Via Electrocardiogram (ECG)
Description: QT interval corrected using the Fridericia formula [QTc (Frid)] - Change from baseline to end of treatment
Time Frame: Baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: msec
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 377 | 364
msec | -0.11 [-1.01 to 0.79] | -0.31 [-1.23 to 0.61]

4. Secondary Outcome: Number of Patients With Shift From Normal to High Rate of Total Ectopic Ventricular Beats as Measured by 24-hour Holter Monitor Assessment
Description: Total ectopic ventricular (VE) beats - number of participants with shift from normal (<50) to high (≥50) from baseline to visit 4.
Time Frame: Baseline and 2 weeks (visit 4)
Population: Data were available for a subset of patients.
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 59 | 63
Participants | 4 | 3

5. Secondary Outcome: Number of Patients With Shift From Normal to High Rate of Total Ectopic Supraventricular Beats as Measured by 24-hour Holter Monitor Assessment
Description: Total ectopic supraventricular (VE) beats - number of participants with shift normal (<50) to high (≥50) from baseline to visit 4.
Time Frame: Baseline and 2 weeks (visit 4)
Population: Data were available for a subset of patients
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 60 | 67
Participants | 4 | 3

6. Secondary Outcome: Total Number of Ventricular Runs as Measured by 24-hour Holter Monitor Assessment
Description: Total ventricular runs - number of participants with shift normal (<1) to high (≥1) from baseline to week 2.
Time Frame: Baseline and 2 weeks (visit 4)
Population: Data were available for a subset of patients.
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 63 | 74
Participants | 2 [13.43 to 18.34] | 1 [8.11 to 13.13]

7. Secondary Outcome: Diary Assessments - Rescue-free Day
Description: Calculated as the number of rescue-free days divided by the number of non missing days in the baseline period times 100%. The results are expressed as the change in % rescue-free days in the baseline period and the active treatment period. A rescue-free day was one in which the patient answered "no" to having used rescue medication that day
Time Frame: baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Rescue Free Day
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 369 | 353
Percentage of Rescue Free Day | 15.88 [13.43 to 18.34] | 10.62 [8.11 to 13.13]

8. Secondary Outcome: Diary Assessments - Symptom-free Day
Description: Calculated as the number of symptom-free days divided by the number of non missing days in the baseline period times 100%. The results are expressed as the change in % symptom-free days in the baseline period and the active treatment period. A symptom-free day was one in which the patient answered "no" to having symptoms that day
Time Frame: baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of Symptom-free day
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 369 | 353
percentage of Symptom-free day | 9.46 [7.55 to 11.37] | 7.58 [5.62 to 9.53]

9. Secondary Outcome: Diary Assessments - Asthma-control Day
Description: Calculated as the number of asthma control days divided by the number of non missing days in the baseline period times 100%. The results are expressed as the change in % asthma control days in the baseline period and the active treatment period. An asthma control day was one in which the patient answered "no" to having symptoms and "0" to the use of rescue medication that day
Time Frame: baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of Asthma-control day
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 369 | 353
percentage of Asthma-control day | 16.68 [14.16 to 19.21] | 11.62 [9.04 to 14.20]

10. Secondary Outcome: Onset of Effect Questionnaire (OEQ)
Description: Number of participants with positive response to Item 2 in questionnaire "During the past week,you could feel your study medication begin to work right away. A positive response was defined as a response of "strongly agree" or "somewhat agree"
Time Frame: 1 week
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 377 | 364
Participants | 172 | 158

11. Secondary Outcome: Onset of Effect Questionnaire (OEQ)
Description: Number of participants with positive response to Item 5 in questionnaire "During the past week, you were satisfied with how quickly you felt your study medication begin to work." The scale was scored on a 5-point Likert scale from strongly agree to strongly disagree. A positive response was defined as a response of "strongly agree" or "somewhat agree"
Time Frame: 1 week
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 377 | 364
Participants | 165 [46.19 to 49.80] | 157 [43.95 to 47.33]

12. Secondary Outcome: Peak Expiratory Flow (PEF) in Morning
Description: Change in AM PEF from baseline (mean over the 2 weeks run-in) to the average of the randomized treatment period.
Time Frame: baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/minute
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 364 | 349
Liters/minute | 30.13 [24.38 to 35.87] | 19.73 [13.86 to 25.59]

13. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: Change in pre-dose FEV1 from baseline (end of run-in, visit 3) to the average of the randomized treatment period
Time Frame: baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 359 | 354
Litres | 0.08 [0.05 to 0.11] | -0.01 [-0.04 to 0.01]

14. Secondary Outcome: Asthma Treatment Satisfaction Measure (ATSM)
Description: Overall score - change from baseline to end of treatment. For 11 individual attributes, expectations were subtracted from the outcomes. This difference and the importance rating were combined in a weighted average which was then multiplied by the raw satisfaction measure. The final derived satisfaction measure was transformed to a 0 to 100 scale, with higher scores representing greater satisfaction.
Time Frame: Baseline and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Symbicort | Budesonide
Number analyzed (Participants) | 203 | 232
units on a scale | 47.99 [46.19 to 49.80] | 45.64 [43.95 to 47.33]

ADVERSE EVENTS:
Arm/Group | Symbicort | Budesonide
Serious Adverse Events (participants affected / at risk) | 12/377 | 15/365
Other Adverse Events (participants affected / at risk) | 98/377 | 84/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=377) | Budesonide (N=365)
Oesophageal Fistula (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia Bacterial (Infections and infestations) | 1 | 1
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body Trauma (Injury, poisoning and procedural complications) | 0 | 1
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Ovarian Mass (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=377) | Budesonide (N=365)
Nasopharyngitis (Infections and infestations) | 26 | 29
Sinusitis (Infections and infestations) | 15 | 23
Viral Upper Respiratory Tract Infection (Infections and infestations) | 22 | 16
Headache (Nervous system disorders) | 36 | 27
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 19 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may use the Multi-Center Study Results and the Site Data for the limited purpose of his or her own research and academic analysis until the earlier of the publication of the first Multi-Center Study at all participating sites